CLINICAL TRIAL: NCT05793450
Title: Pharmacokinetics of IBI362 in Subjects With and Without Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CIBI362D102
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — mazdutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IBI362 - Mild and Moderate Renal Impairment (Experimental): Group 2 - IBI362 administered SC to participants with mild and moderate renal impairment.
  Interventions: Drug: IBI362
- IBI362 - Healthy (Experimental): Group 1 - IBI362 administered subcutaneously (SC) to healthy participants with normal renal function.
  Interventions: Drug: IBI362
- IBI362 - Severe Renal Impairment (Experimental): Group 3 - IBI362 administered SC to participants with severe renal impairment.
  Interventions: Drug: IBI362

INTERVENTIONS:
Drug: IBI362 — 2.0mg, SC, single dose

SUMMARY:
The purpose of this study is to assess how fast IBI362 gets into the blood stream and how long it takes the body to remove it in participants with impaired kidney function compared to healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* All Participants:

  o The weight of male subjects is not less than 50 kg, and the body weight of female subjects is not less than 45 kg, and the body mass index (BMI) is within the range of 20~30 kilograms per meter squared (kg/m²), inclusive, at screening
* Healthy Participants:

  -- Healthy males or females as determined by medical history, physical examination, and other screening procedures, with normal renal function, assessed by estimated glomerular filtration rate (eGFR) ≥90 milliliters per minute (mL/min) at screening
* Participants with Renal Impairment:

  * Males or females with stable mild to severe renal impairment, assessed by eGFR

Exclusion Criteria:

* All Participants:

  * Pregnant or lactating women, or men or women who are of childbearing potential and are not willing to use contraception within 6 months from the screening period to the administration of the study drug
  * Have known allergies to IBI362 or related compounds
  * Have a personal or family history of medullary thyroid carcinoma or have multiple endocrine neoplasia syndrome type 2
  * Have serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5× the upper limit of normal (ULN) or total bilirubin (TBL) >1× ULN
  * Severe gastrointestinal diseases (such as active ulcer, pyloric obstruction, inflammatory bowel disease, etc.) occurred within 6 months before screening, or received gastrointestinal surgery or long-term use of drugs that directly affect gastrointestinal motility due to chronic gastrointestinal diseases
  * Have a history of acute and chronic pancreatitis, or serum amylase and/or lipase ≥ 1.5× ULN at screening, or fasting Triglyceride ≥ 5.64 mmol/L (500 mg/dl)
* Participants with Renal Impairment:

  * obstructive urinary tract diseases (such as urinary stones, urinary tract obstruction caused by abdominal space-occupying lesions, etc.) or renal dysfunction caused by special types of renal parenchymal damage (such as polycystic kidney, medullary sponge kidney, Renal tumors, etc.) and/or patients with renal impairment who have diseases that are not related to renal disease but can cause renal impairment (eg, renal artery stenosis, acute drug injury, severe infection, hypovolemia, heart failure, etc.).
  * Have a history of kidney transplant
  * The treatment medication and/or the treatment medication of other comorbid diseases have been taken stably for less than 1 month at screening, or there are new medications within 1 month before screening (except temporary or intermittent use of drugs, such as Erythropoietin once a month, or diuretics as needed, etc.), or received any drug known to alter renal tubular creatinine secretion within 14 days or 5 half-lives before screening, such as cimetidine D, trimethoprim or cibenzoline, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of IBI362 | Predose through 1344 hours postdose
PK: Area Under the Concentration Versus Time Curve (AUC) of IBI362 | Predose through 1344 hours postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Aerospace Center Hospital, Beijing, Beijing Municipality, China